CLINICAL TRIAL: NCT05005416
Title: Efficacy of a Culturally Adapted Cognitive Behavioral Based Physical Therapy Intervention for Latinos With Chronic Spine Pain
Brief Title: Goal Oriented Activity for Latinos With Spine Pain
Acronym: GOALS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH); Family Health Centers of San Diego (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 228489; U54MD012397 (NIH)
Record Dates: First submitted 2021-08-05; First posted 2021-08-13 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Low Back Pain; Neck Pain; Chronic Pain; Chronic Low-back Pain
Keywords: physical therapy; rehabilitation; cognitive behavioral; hispanic; health disparities; telehealth
MeSH Terms: conditions — Low Back Pain; Neck Pain; Chronic Pain

STUDY DESIGN:
Intervention Model Description: The primary purpose of this interventional study is to determine the efficacy of a culturally adapted cognitive behavioral based tele-rehabilitation program compared to usual care for Hispanics/Latinos with chronic neck or low back pain. The main objective of the GOALS intervention is to improve pain-related disability in Hispanics/Latinos with chronic spine pain. The interventional study model is a single site, 2-arm parallel assignment randomized clinical trial with blinded assessors. After completing the baseline assessment, enrolled participants will be stratified by sex (male, female) and diagnosis (low back pain/neck pain) and randomized into either the GOALS intervention arm or the Usual Care control arm.
Who Masked: Outcomes Assessor
Masking Description: Research assistants conducting all assessments and biostatisticians conducting the analyses will be masked to treatment group. Participants, physical therapist providers, investigators, recruitment coordinators, and project managers will not be masked. Physical therapists who provide the Usual Care intervention will be naïve to the purpose of the study and details of the GOALS intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GOALS Intervention (Experimental): The experimental arm is an 8-week cognitive-behavioral based physical therapy (PT) intervention for chronic spine pain. The manualized intervention utilizes a hybrid tele-rehabilitation delivery model. GOALS comprises an initial in-person evaluation (60 min) by a research physical therapist, followed by 6 remote treatment sessions (30-45 min each) conducted by the same physical therapist once a week by telephone. A second in-person evaluation is conducted at the midpoint of the GOALS intervention to assess progress and advance the participant's home exercise program.
  Interventions: Behavioral: GOALS Intervention
- Usual Care Physical Therapy (Active Comparator): The control arm is Usual Care physical therapy (PT) at a local Federally Qualified Health Center (FQHC), which offers PT services at 4 outpatient clinics across San Diego county. Participants in the Usual Care group attend an initial PT evaluation at a FQHC Physical Rehabilitation Clinic. The frequency and type of PT intervention are then determined by the treating physical therapist in accordance with standard clinical practice at the FQHC.
  Interventions: Behavioral: Usual Care Physical Therapy

INTERVENTIONS:
Behavioral: GOALS Intervention — Weekly treatment sessions are comprised of a graded activity program focused on goal setting in 4 treatment domains: therapeutic exercise, aerobic activity, functional activity, and pain coping skills. Instruction in cognitive behavioral coping skills for pain include: explaining pain (pain neuroscience education), pacing, soliciting positive social support, cognitive restructuring, present mindedness, and symptom self-management planning.
  Arms: GOALS Intervention
Behavioral: Usual Care Physical Therapy — Usual care will be characterized by extracting the following variables from participants' electronic health record: date of physician referral to physical therapy for neck or low back pain diagnosis (index referral), attendance of at least one PT visit (adherence), dates of first and last PT visits for index referral (duration of care), number of PT visits attended across an 8-week episode of care for the index referral (number of visits), clinic where PT services were provided (service location), and CPT billing codes issued during the episode of care for the index referral (type and frequency of treatments provided).
  Arms: Usual Care Physical Therapy

SUMMARY:
The primary purpose of the study is to determine the efficacy of a culturally adapted cognitive behavioral based tele-rehabilitation program compared to usual care for Hispanics/Latinos with chronic neck or low back pain. Goal Oriented Activity for Latinos with Spine Pain (GOALS) is an evidence-based cognitive behavioral physical therapy program that has been adapted for Hispanics/Latinos with chronic spine pain. GOALS combines 2 in-person evaluation sessions with 6 telephone treatment sessions provided once a week for 8 weeks by a physical therapist trained in cognitive behavioral approaches for pain management. Usual Care involves 8 weeks of in-person treatment as recommended by a physical therapist at a Federally Qualified Health Center (FQHC) outpatient rehabilitation clinic. The primary outcome that will be evaluated is pain-related disability as measured by the Brief Pain Inventory Pain Interference scale. It is hypothesized that participants in the GOALS intervention will experience a greater improvement in pain-related disability than participants in the Usual Care group.

DETAILED DESCRIPTION:
123 Hispanics/Latinos with chronic spine pain will be identified through consecutive sampling of patients at a local FQHC who were referred by their primary care physician to physical therapy (PT) for neck or low back pain. Participants who are deemed eligible and enroll in the study will be scheduled for the first study assessment, where they will provide written informed consent for participation. Participation includes 4 study assessments and 8-weeks of treatment with either GOALS or Usual Care PT. Participants will be stratified by sex (male/female) and diagnosis (low back pain/neck pain) and randomized into either the GOALS or the Usual Care group following completion of the Baseline assessment. Study assessments will be conducted 1-week before (Baseline) and 1-week (Post), 3-months (3-mo Post), and 6-months (6-mo Post) after completing 8 weeks of GOALS or Usual Care PT.

The projected sample size for GOALS changed from N=138 to N=123 after adding an eligibility criterion requiring participants to attend the PT evaluation. Our power analysis indicated N=98 participants is the smallest sample size needed to detect the effect of the GOALS intervention. Before beginning the trial, we estimated a 41% attrition rate given data from the partnering clinic, suggesting we needed to recruit N=138 to meet our N=98 sample size. However, we added an inclusion criterion that participants need to attend the initial PT evaluation in order to be enrolled in the study. We retained an estimated attrition rate of 20% of enrolled participants, requiring an initial sample size of N=123 to meet the N=98 minimum sample size.

The primary aim of the study is to determine the efficacy of a culturally adapted cognitive behavioral based PT tele-rehabilitation program compared to usual care in Hispanics/Latinos with chronic spine pain, based on improvement in the pain interference scale in the Brief Pain Inventory after treatment (primary outcome). The 1-week post-intervention assessment will be analyzed using a linear regression model. The time by condition (GOALS vs. Usual Care) interaction term will be added to the models to assess for intervention effects. If the interaction is not significant, the main effect for time and condition will be assessed. For all outcomes, the models will be adjusted for sociodemographic and clinical characteristics that may affect treatment response. Secondary outcomes of pain interference at other time-points (3- and 6-mo Post) and patient reported outcomes and physical performance measures at all time points will be evaluated in the same manner. It is hypothesize that participation in the GOALS intervention compared to Usual Care will result in greater improvements in pain interference (primary outcome), as well as secondary patient reported outcomes and physical performance measures.

Pre-planned secondary analyses will explore biological/physical, psychological, and environmental moderators and mediators of treatment response. The dependent variable for this analysis will be treatment response, whereby participants will be dichotomized into responder and non-responder groups based on a ≥30% reduction in pain interference as recommended by IMMPACT guidelines. An exploratory, backward selection approach using separate multivariate logistic regression models will be used to identify predictors that are most strongly related to treatment response. These variables will then be entered into a single combined multivariate logistic regression model adjusted for sociodemographic covariates of treatment response. The study will also explore potential mediators of treatment response with structural equation modeling (SEM) using maximum likelihood estimation methods. Parameter estimates will be evaluated and indirect effects, reflecting mediation, will be calculated and examined for statistical significance and clinical meaningfulness. It is hypothesized that baseline indicators for high fear of movement and sedentary behavior will predict a positive response to the GOALS intervention. However, the study will also collect and analyze other candidate predictors of treatment response based on a conceptual model of the pain experience in Hispanics/Latinos.

ELIGIBILITY:
Inclusion Criteria:

* Referred to physical therapy by primary care physician
* 18-66 years old
* Hispanic
* Diagnosis of chronic neck or low back pain
* Must attend at least 1 physical therapy treatment session

Exclusion Criteria:

* Tumor, infection, or other major medical problem affecting the neck or low back
* Health problems that severely affect ability to move, walk one block, or participate in exercise
* Presence of external incentives for non-recovery (e.g., litigation, worker's compensation benefits)
* Initiating or receiving any new psychotherapy or behavioral health treatment for the neck or low back pain during the observation period
* Diagnosis of a major psychological condition (e.g., schizophrenia, psychosis, bipolar disorder)
* Inability to provide a stable address with access to a telephone or any other reason that would preclude participation in a telephone-based intervention
* Cohabitating with a GOALS/Metas participant
* Pregnant or lactating

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2021-08-04 (Actual); Primary Completion 2024-07-23 (Actual); Study Completion 2024-12-16 (Actual)

PRIMARY OUTCOMES:
Brief Pain Inventory (BPI) - Pain Interference | Change from Baseline to Post-Intervention (1-week)
  To assess global pain-related disability. Scale values: 0 (min) to 10 (max). Decreases in score indicate improvement in outcomes.

SECONDARY OUTCOMES:
Brief Pain Inventory (BPI) - Pain Interference | Change from Baseline to Post-Intervention (3-month, 6-month)
  To assess global pain-related disability. Scale values: 0 (min) to 10 (max). Decrease in score indicate improvement in outcomes.
Brief Pain Inventory (BPI) - Pain Intensity | Change from Baseline to Post-Intervention (1-week, 3-month, 6-month)
  To assess global pain severity. Scale values: 0 (min) to 10 (max). Decrease in score indicate improvement in outcomes.
PEG-3 | Change from Baseline to Post-Intervention (1-week, 3-month, 6-month)
  To assess global pain intensity and pain interference. Scale values: 0 (min) to 10 (max). Decrease in score indicate improvement in outcomes.
Neck Disability Index (NDI) | Change from Baseline to Post-Intervention (1-week, 3-month, 6-month)
  To assess regional pain-related disability for people with neck pain. Scale values: 0% (min) to 100% (max). Decrease in score indicate improvement in outcomes.
Modified Oswestry Disability Index (ODI) | Change from Baseline to Post-Intervention (1-week, 3-month, 6-month)
  To assess regional pain-related disability for people with low back pain. Scale values: 0% (min) too 100% (max). Decrease in score indicate improvement in outcomes.
Patient Specific Functional Scale (PSFS) | Change from Baseline to Post-Intervention (1-week, 3-month, 6-month)
  To assess ability to perform patient-identified functional activities. Scale values: 0 (min) to 10 (max). Increase in score indicate improvement in outcomes.
6-Meter Walk Test | Change from Baseline to Post-Intervention (1-week)
  To assess preferred and maximum gait speeds. Scale is measured in seconds. Decrease in score indicate improvement in outcomes.
30-s Sit-to-Stand | Change from Baseline to Post-Intervention (1-week)
  To assess number of repetitions for a sit-to-stand functional performance task for people with low back pain. Scale is measured in number of repetitions. Increase in score indicates improvement in outcomes.

OTHER OUTCOMES:
Treatment Expectancy Measure | Baseline
  To assess participant expectancy related to treatment condition assigned. Scale values: 0 (min) to 10 (max). Higher scores indicate better therapeutic alliance.
Kim Alliance Scale (KAS) | Post-Intervention (1-week)
  To assess therapeutic alliance for the treatment condition rendered. Scale values: 16 (min) to 64 (max). Higher scores indicate better therapeutic alliance.
Global Impression of Change (GIC) | Post-Intervention (1-week, 3-month, 6-month)
  To assess self-reported improvement with intervention. Scale values: 1 (min) to 7 (max). Lower scores indicate better outcomes.
Global Rating of Satisfaction (GRS) | Post-Intervention (1-week, 3-month, 6-month)
  To assess self-reported satisfaction with intervention. Scale values: 1 (min) to 7 (max). Lower scores indicate better outcomes.
Fear Avoidance Beliefs Questionnaire (FABQ) | Baseline; Post Intervention (1-week, 3-month)
  To assess fear of movement associated with neck or low back pain. Physical activity subscale: Scale values: 0 (min) to 24 (max). Work Subscale: Scale values: 0 (min) to 42 (max). Decrease in scores indicate improvement in outcomes.
Pain Catastrophizing Scale (PCS) | Baseline; Post-Intervention (1-week, 3-month)
  To assess pain catastrophizing. Scale values: 0 (min) to 52 (max). Decrease in scores indicate improvement in outcomes.
Medical Outcomes Study - Social Support Measure (MOS-SS) | Baseline; Post-Intervention (1-week)
  To assess social support. Scale values: 0% (min) to 100% (max). Increase in scores indicate improvement in outcomes.
New General Self-Efficacy Scale (GSES) | Baseline; Post-Intervention (1-week, 3-month)
  To assess general self-efficacy. Scale values: 1 (min) to 5 (max). Increase in scores indicate an improvement in outcomes.
Pain Self-Efficacy Questionnaire (PSEQ) | Baseline; Post-Intervention (1-week, 3-month)
  To assess self-efficacy specifically related to pain. Scale values: 0 (min) to 60 (max). Increase in scores indicate improvement in outcomes.
PROMIS Short-Form Anxiety 4a | Baseline; Post-Intervention (1-week, 3-month)
  To assess generalized anxiety. Scale values: 0 (min) to 100 (max). Decrease in scores indicate improvement in outcomes.
PROMIS Short-Form Depression 4a | Baseline; Post-Intervention (1-week, 3-month)
  To assess depressive symptoms. Scale values: 0 (min) to 100 (max). Decrease in scores indicate improvement in outcomes.
PROMIS Short-Form Sleep Disturbance | Baseline; Post-Intervention (1-week, 3-month)
  To assess sleep disturbance. Scale values: 0 (min) to 100 (max). Decrease in scores indicate improvement in outcomes.
PROMIS Short-Form Physical Function 4a | Baseline, Post-Intervention (1-week, 3-month)
  To assess generalized physical function. Scale values: 0 (min) to 100 (max). Increase in scores indicate improvement in outcomes.
PROMIS Short-Form Ability to Participate 4a | Baseline; Post-Intervention (1-week, 3-month)
  To assess participation in social roles and activities. Scale values: 0 (min) to 100 (max). Increase in scores indicate improvement in outcomes.
Rapid Assessment of Physical Activity (RAPA) Aerobic | Baseline; Post-Intervention (1-week, 3-month)
  To assess self-reported physical activity. Aerobic scale values: 1 (min) to 7 (max). Increase in scores indicate improvement in outcomes.
Rapid Assessment of Physical Activity (RAPA) Strength and Flexibility | Baseline; Post-Intervention (1-week, 3-month)
  To assess self-reported physical activity. Strength & Flexibility scale values: 0 (min) to 3 (max). Increase in scores indicate improvement in outcomes.
Self-Efficacy and Exercise Habits Survey (SEHS) | Baseline; Post-Intervention (1-week, 3-month)
  To assess self-efficacy specifically related to exercise. Scale values: 1 (min) to 5 (max). Increase in scores indicate improvement in outcomes.
Physical Activity (Actigraph) | Baseline; Post-Intervention (1-week)
  Objective measure of physical activity. Physical activity scale values: 0% (min) to 100% (max) (increase in score indicate improvement in outcomes.)
Physical Activity and Sedentary Behavior (Actigraph) | Baseline; Post-Intervention (1-week)
  Objective measures of physical activity. Sedentary behavior scale values: 0% (min) to 100% (max) (decrease in score indicate improvement in outcomes.)
Sleep Efficiency (Actigraph) | Baseline; Post-Intervention (1-week)
  Objective measure of sleep behavior. Efficiency 0-100% (increase is an improvement).
Sleep Duration (Actigraph) | Baseline; Post-Intervention (1-week)
  Objective measure of sleep behavior. Time Asleep in minutes (increase is an improvement).
Sleep Onset (Actigraph) | Baseline; Post-Intervention (1-week)
  Objective measure of sleep behavior. Sleep Onset Latency in minutes (decrease is an improvement).
Posture and Movement Measures (DorsaVi) | Baseline; Post-Intervention (1-week)
  To assess spine posture and movement and associated pain behavior during clinical tests and daily activities.
Goal Attainment Scale | Once weekly during 8-week GOALS intervention
  To assess the extent to which participants attain weekly goals in the GOALS intervention. Scale values: -2 (min) to 2 (max). Higher scores indicate greater adherence to weekly goals.
Adverse Event Checklist | Once weekly during 8-week GOALS intervention
  To assess type and frequency of treatment-related adverse events.
Post-Intervention Survey | Post-Intervention (3-month, 6-month)
  To assess the extent to which participants are continuing to utilize the GOALS/Metas program activities and the importance of the physical therapy treatment in management of their chronic spine pain.

CONTACTS AND LOCATIONS:
Overall Officials: Katrina Monroe, PT, Ph.D, Principal Investigator — San Diego State University; Sara Gombatto, PT, Ph.D, Principal Investigator — San Diego State University
Locations (2):
- United States (2):
  - Family Health Centers of San Diego, San Diego, California
  - SDSU HealthLINK Center, San Diego, California

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (including data dictionaries) that underlie the results reported in publications, after deidentification (text, tables, figures, appendices), will be available. Other documents that will be made available include: Study Protocol, Statistical Analysis Plan, Analytic Code, Informed Consent Form, Patient Guide (English/Spanish), and Therapist Guide (English/Spanish). Data will be available for individual participant data meta-analysis beginning 6 months and ending 5 years following article publication.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Beginning 6 months and ending 5 years following article publication.
Access Criteria: Data will be available to investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose by the San Diego State University HealthLINK Advisory Board. To gain access, data requestors will need to sign a data access agreement. Proposals should be directed to sgombatto@sdsu.edu. Data are available for 5 years through the San Diego State University HealthLINK Health Science Knowledge Repository website.

REFERENCES:
- [Background] Archer KR, Devin CJ, Vanston SW, Koyama T, Phillips SE, Mathis SL, George SZ, McGirt MJ, Spengler DM, Aaronson OS, Cheng JS, Wegener ST. Cognitive-Behavioral-Based Physical Therapy for Patients With Chronic Pain Undergoing Lumbar Spine Surgery: A Randomized Controlled Trial. J Pain. 2016 Jan;17(1):76-89. doi: 10.1016/j.jpain.2015.09.013. Epub 2015 Oct 23. PMID 26476267
- [Background] Archer KR, Motzny N, Abraham CM, Yaffe D, Seebach CL, Devin CJ, Spengler DM, McGirt MJ, Aaronson OS, Cheng JS, Wegener ST. Cognitive-behavioral-based physical therapy to improve surgical spine outcomes: a case series. Phys Ther. 2013 Aug;93(8):1130-9. doi: 10.2522/ptj.20120426. Epub 2013 Apr 18. PMID 23599351
- [Background] Bennell KL, Ahamed Y, Jull G, Bryant C, Hunt MA, Forbes AB, Kasza J, Akram M, Metcalf B, Harris A, Egerton T, Kenardy JA, Nicholas MK, Keefe FJ. Physical Therapist-Delivered Pain Coping Skills Training and Exercise for Knee Osteoarthritis: Randomized Controlled Trial. Arthritis Care Res (Hoboken). 2016 May;68(5):590-602. doi: 10.1002/acr.22744. PMID 26417720
- [Background] da C Menezes Costa L, Maher CG, Hancock MJ, McAuley JH, Herbert RD, Costa LO. The prognosis of acute and persistent low-back pain: a meta-analysis. CMAJ. 2012 Aug 7;184(11):E613-24. doi: 10.1503/cmaj.111271. Epub 2012 May 14. PMID 22586331
- [Background] Mackey S. National Pain Strategy Task Force: the strategic plan for the IOM Pain Report. Pain Med. 2014 Jul;15(7):1070-1. doi: 10.1111/pme.12490. No abstract available. PMID 25059928
- [Background] Gagnon CM, Matsuura JT, Smith CC, Stanos SP. Ethnicity and interdisciplinary pain treatment. Pain Pract. 2014 Jul;14(6):532-40. doi: 10.1111/papr.12102. Epub 2013 Jul 29. PMID 23889982
- [Background] Hogg-Johnson S, van der Velde G, Carroll LJ, Holm LW, Cassidy JD, Guzman J, Cote P, Haldeman S, Ammendolia C, Carragee E, Hurwitz E, Nordin M, Peloso P; Bone and Joint Decade 2000-2010 Task Force on Neck Pain and Its Associated Disorders. The burden and determinants of neck pain in the general population: results of the Bone and Joint Decade 2000-2010 Task Force on Neck Pain and Its Associated Disorders. Spine (Phila Pa 1976). 2008 Feb 15;33(4 Suppl):S39-51. doi: 10.1097/BRS.0b013e31816454c8. PMID 18204398
- [Background] Hollingshead NA, Ashburn-Nardo L, Stewart JC, Hirsh AT. The Pain Experience of Hispanic Americans: A Critical Literature Review and Conceptual Model. J Pain. 2016 May;17(5):513-28. doi: 10.1016/j.jpain.2015.10.022. Epub 2016 Jan 30. PMID 26831836
- [Background] Hoy D, March L, Brooks P, Blyth F, Woolf A, Bain C, Williams G, Smith E, Vos T, Barendregt J, Murray C, Burstein R, Buchbinder R. The global burden of low back pain: estimates from the Global Burden of Disease 2010 study. Ann Rheum Dis. 2014 Jun;73(6):968-74. doi: 10.1136/annrheumdis-2013-204428. Epub 2014 Mar 24. PMID 24665116
- [Background] Hoy D, March L, Woolf A, Blyth F, Brooks P, Smith E, Vos T, Barendregt J, Blore J, Murray C, Burstein R, Buchbinder R. The global burden of neck pain: estimates from the global burden of disease 2010 study. Ann Rheum Dis. 2014 Jul;73(7):1309-15. doi: 10.1136/annrheumdis-2013-204431. Epub 2014 Jan 30. PMID 24482302
- [Background] Kamper SJ, Apeldoorn AT, Chiarotto A, Smeets RJ, Ostelo RW, Guzman J, van Tulder MW. Multidisciplinary biopsychosocial rehabilitation for chronic low back pain. Cochrane Database Syst Rev. 2014 Sep 2;2014(9):CD000963. doi: 10.1002/14651858.CD000963.pub3. PMID 25180773
- [Background] Katz JN. Lumbar disc disorders and low-back pain: socioeconomic factors and consequences. J Bone Joint Surg Am. 2006 Apr;88 Suppl 2:21-4. doi: 10.2106/JBJS.E.01273. PMID 16595438
- [Background] Nielsen M, Keefe FJ, Bennell K, Jull GA. Physical therapist-delivered cognitive-behavioral therapy: a qualitative study of physical therapists' perceptions and experiences. Phys Ther. 2014 Feb;94(2):197-209. doi: 10.2522/ptj.20130047. Epub 2013 Sep 12. PMID 24029300
- [Background] Plesh O, Adams SH, Gansky SA. Racial/Ethnic and gender prevalences in reported common pains in a national sample. J Orofac Pain. 2011 Winter;25(1):25-31. PMID 21359234
- [Background] Rahim-Williams B, Riley JL 3rd, Williams AK, Fillingim RB. A quantitative review of ethnic group differences in experimental pain response: do biology, psychology, and culture matter? Pain Med. 2012 Apr;13(4):522-40. doi: 10.1111/j.1526-4637.2012.01336.x. Epub 2012 Mar 5. PMID 22390201
- [Background] Cote P, Cassidy DJ, Carroll LJ, Kristman V. The annual incidence and course of neck pain in the general population: a population-based cohort study. Pain. 2004 Dec;112(3):267-273. doi: 10.1016/j.pain.2004.09.004. PMID 15561381
- [Background] Stewart WF, Ricci JA, Chee E, Morganstein D, Lipton R. Lost productive time and cost due to common pain conditions in the US workforce. JAMA. 2003 Nov 12;290(18):2443-54. doi: 10.1001/jama.290.18.2443. PMID 14612481
- [Background] Turner JA, Mancl L, Aaron LA. Short- and long-term efficacy of brief cognitive-behavioral therapy for patients with chronic temporomandibular disorder pain: a randomized, controlled trial. Pain. 2006 Apr;121(3):181-194. doi: 10.1016/j.pain.2005.11.017. Epub 2006 Feb 21. PMID 16495014
- [Background] Woods MP, Asmundson GJG. Evaluating the efficacy of graded in vivo exposure for the treatment of fear in patients with chronic back pain: a randomized controlled clinical trial. Pain. 2008 Jun;136(3):271-280. doi: 10.1016/j.pain.2007.06.037. Epub 2007 Aug 22. PMID 17716819
- [Background] Zettel-Watson L, Rutledge DN, Aquino JK, Cantero P, Espinoza A, Leal F, Jones CJ. Typology of chronic pain among overweight Mexican Americans. J Health Care Poor Underserved. 2011 Aug;22(3):1030-47. doi: 10.1353/hpu.2011.0092. PMID 21841294
- [Background] Van Dyke BP, Newman AK, Morais CA, Burns JW, Eyer JC, Thorn BE. Heterogeneity of Treatment Effects in a Randomized Trial of Literacy-Adapted Group Cognitive-Behavioral Therapy, Pain Psychoeducation, and Usual Medical Care for Multiply Disadvantaged Patients With Chronic Pain. J Pain. 2019 Oct;20(10):1236-1248. doi: 10.1016/j.jpain.2019.04.006. Epub 2019 Apr 22. PMID 31022555
- [Derived] Gombatto SP, Archer KR, Wegener ST, Hernandez Y, Lin SF, Godino J, Van Dyke J, Liu J, Monroe KS. Protocol for a Parallel Group Randomized Clinical Trial Comparing a Culturally Adapted Cognitive Behavioral Telerehabilitation Intervention to Usual Physical Therapy for Latino Patients With Chronic Spine Pain. Phys Ther. 2023 Sep 1;103(9):pzad068. doi: 10.1093/ptj/pzad068. PMID 37364033

DOCUMENTS (1):
  • Informed Consent Form (2023-08-10): https://cdn.clinicaltrials.gov/large-docs/16/NCT05005416/ICF_000.pdf